CLINICAL TRIAL: NCT03355508
Title: Impact of the Arteriovenous Fistula Puncture Technique On the Hemodialysis Session For Patient and Caregiver
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poissy-Saint Germain Hospital (Other)
Responsible Party: Principal Investigator, Valérie LOIZEAU, Impact of the Arteriovenous Fistula Puncture Technique On the Hemodialysis Session For Patient and Caregiver, Poissy-Saint Germain Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: TECHFAVHEMO
Record Dates: First submitted 2017-10-25; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Arterio-venous Fistula, Puncture, Chronic Desease
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- puncture bevel up (Other)
  Interventions: Device: pucture in the arteriovenous fistula
- puncture bevel domn (Other)
  Interventions: Device: pucture in the arteriovenous fistula

INTERVENTIONS:
Device: pucture in the arteriovenous fistula — The compression time will be measured with a stopwatch so that it is objective and accurate, although the compression times range from minute to minute.
  An initial 2-week observation phase (phase 1) will establish a reference time for each patient using the most common puncture technique in the department: bevel up.
  We will evaluate the patient's reference time by counting the time of compression using a stopwatch for 2 weeks (ie 6 sessions) and we will take an average.
  A draw will determine for each patient the order in which the direction of the needles will be used.
  After this determination of the reference time, the patient will enter two successive phases where it will be punctured bevel up (phase 2) and then down (phase 3) or vice versa following the draw.

SUMMARY:
40000 patients are hemodialysis each year in France .

In the case of chronic care, 78% of patients have an arteriovenous fistula. In order to perform the hemodialysis session, 2 techniques of puncture of the fistula are possible:

* Bevel puncture upwards then flipping the needle
* or puncture bevel down. At present, there is no consensus or study on the technique of puncture fistula which generates different professional practices.

ELIGIBILITY:
Inclusion Criteria:

* Patient in chronic renal failure treated by hemodialysis with native arteriovenous fistula as a vascular approach.
* Adult of age and sex indifferent.
* Normal puncture of the fistula with two needles (bipuncture).
* Fistula use for more than 3 months.
* Beneficiary of Medicare or State Medical Aid.
* No opposition to participation in the study.

Exclusion Criteria:

* Patient who does not speak and does not understand French.
* Hemodialysis patient awaiting a transplant by a living donor.
* Patient with more than 2 AVF dilatations in the last 6 months.
* Patient with prosthetic arteriovenous fistula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Compression time required for hemostasis | period of 3 weeks
  The primary endpoint is the compression time required for hemostasis after needle removal, which is stable over a 3-week period.
  The compression time will be measured with a stopwatch so that it is objective and accurate, although the compression times range from minute to minute. An initial 2-week observation phase (phase 1) will establish a reference time for each patient using the most common puncture technique in the department: bevel up. We will evaluate the patient's reference time by counting the time of compression using a stopwatch for 2 weeks (ie 6 sessions) and we will take an average. A draw will determine for each patient the order in which the direction of the needles will be used. After this determination of the reference time, the patient will enter two successive phases where it will be tapped bevel up (phase 2) and then down (phase 3) or vice versa following the draw.

CONTACTS AND LOCATIONS:
Locations (1):
- CH Poissy st Germain, Poissy, France